CLINICAL TRIAL: NCT01430715
Title: Active Video Gaming Compared to Unstructured, Outdoor Play in Children: Measurements of Estimated Energy Expenditure and Measured Percent Time in Moderate-to-Vigorous Physical Activity
Brief Title: Estimating Energy Expenditure in Active Video Gaming Compared to Unstructured, Outdoor Play in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 8556
Record Dates: First submitted 2011-08-05; First posted 2011-09-08 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Motor Activity
Keywords: active video game; video gaming; accelerometery; MVPA; outdoor play; children; unstructured; energy expenditure
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Outside play (Experimental)
  Interventions: Other: Active vido games and outdoor play
- Active video game (Experimental)
  Interventions: Other: Active vido games and outdoor play

INTERVENTIONS:
Other: Active vido games and outdoor play — Fifteen children, aged 5- to 8- years, attending a nearby preschool, with a normal body mass index (BMI)-for-age percentile between, > 5th % to < 85th %.BMI, will participate in unstructured, outdoor play and one AVGs in a randomized order. Activity type, duration and intensity will be measured via accelerometery and direct observation. The energy expenditure (EE) will be calculated from Metabolic Equivalent (MET) values and the percent of time each activity meets MVPA intensity will be calculated. A MET is the energy cost of the activity expressed as kilocalories expended per kilogram of body weight per hour of activity. If EE and intensity in AVG play is similar to EE and intensity in outdoor play, then AVG play could be a great supplement to efforts aimed at increasing PA in children.
  Other Names: active video games; outdoor play; accelerometery

SUMMARY:
The increasing use of sedentary screen-based activities (SBAs) has been most recently blamed for children and adolescents' lack of engagement in physical activity (PA). Studies indicate a large portion of children participate high-levels of sedentary SBAs and the sedentary SBAs appear to compete for time to engage in PA. If sedentary behavior is a substitute for PA, to help increase PA, strategies need to be put into place that helps to decrease sedentary behaviors.

One modification to sedentary videogames that may increase PA in children is to alter sedentary videogames so that the videogames actually provide an option to engage in PA, rather than to be sedentary. These types of games then don't compete with PA, but actually are a source of PA. These types of videogames are called active video games (AVG) or "Exer-gaming." Previous research demonstrates that energy-expenditure (EE) in AVG play is comparable to moderate-intensity walking and produce greater EE than sedentary SBAs. However, previous studies have been limited to measuring EE in AVG play to walking either on a treadmill or in a structured setting. Studies have not investigated the EE of AVG play compared to the EE in free-living outdoor play. Thus, the purpose of the proposed study is to determine whether a greater EE is released during AVG play compared to free-living, outdoor play in children.

DETAILED DESCRIPTION:
Fifteen children, aged 5- to 8- years, attending a nearby preschool, with a normal body mass index (BMI)-for-age percentile between, > 5th % to < 85th %.BMI, will participate in unstructured, outdoor play and one AVGs in a randomized order. Activity type, duration and intensity will be measured via accelerometery and direct observation. The EE will be calculated from Metabolic Equivalent (MET) values and the percent of time each activity meets MVPA intensity will be calculated. A MET is the energy cost of the activity expressed as kilocalories expended per kilogram of body weight per hour of activity (7). If EE and intensity in AVG play is similar to EE and intensity in outdoor play, then AVG play could be a great supplement to efforts aimed at increasing PA in children.

Specific Aims:

1. To measure the EE acquired in 15 minutes during an AVG, an adventure game, as compared to unstructured outdoor play in children 5- to 8- years of age.
2. To compare the percent of time each activity meets the definition of MVPA (MET value >3) in children aged 5- to 8-years of age.

ELIGIBILITY:
Inclusion Criteria:

* All children between 5- to 8- years of age and enrolled in the ELC, with parental consent can participate. Children must be healthy, with an absence of any known cardiopulmonary, metabolic, or orthopedic disease condition or ailment that would limit their participation in the study. Also, children with any type of grass allergy and sensitivity to sunlight will not be included in the study. Additionally, children must be of healthy weight with a body mass index (BMI)-for-age percentile between, > 5th % to < 85th %. Eligible children must also agree to be observed during outdoor activity and while playing the video game.

Exclusion Criteria:

* Children who are not between 5- to 8- years of age and those who are not enrolled in the ELC, and do not obtain parental consent will not be allowed to participate. Children must be healthy, those with any known cardiopulmonary, metabolic, or orthopedic disease condition or aliment that would limit their physical activity, cannot participate in the study. Also, children with any type of grass allergy and sensitivity to sunlight will not be included in the study. Additionally, children must be of healthy weight with a body mass index (BMI)-for-age percentile between, > 5% to < 85%. Children above or below the healthy weight criteria (body mass index (BMI)-for-age percentile below the 5th percentile or above the 85th percentile), will be ineligible and not be able to participate in the study. Eligible children must also agree to be observed during outdoor activity and video-recorded while playing the video game, those children who do not agree to be observed cannot participate in the research study.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Measured the EE acquired in 15 minutes during an AVG, an adventure game, as compared to unstructured outdoor play in children 5- to 8- years of age | within the study's 4 month period
  Fifteen children, aged 5- to 8- years, with a normal body mass index (BMI)-for-age, will participate in unstructured, outdoor play and one AVGs in a randomized order. Activity type, duration and intensity will be measured via accelerometery and direct observation. The energy expenditure (EE) will be calculated from Metabolic Equivalent (MET) values and the percent of time each activity meets MVPA intensity will be calculated. If EE and intensity in AVG play is similar to EE and intensity in outdoor play, then AVG play could be a great supplement to efforts aimed at increasing PA in children.

SECONDARY OUTCOMES:
Compared the percent of time each activity meets the definition of MVPA (MET value >3) in children aged 5- to 8-years of age | within the study's 4 month time frame
  Fifteen children, aged 5- to 8- years, with a normal body mass index (BMI)-for-age, will participate in unstructured, outdoor play and one AVGs in a randomized order. Activity type, duration and intensity will be measured via accelerometery and direct observation. The energy expenditure (EE) will be calculated from Metabolic Equivalent (MET) values and the percent of time each activity meets MVPA intensity will be calculated. If EE and intensity in AVG play is similar to EE and intensity in outdoor play, then AVG play could be a great supplement to efforts aimed at increasing PA in children.

CONTACTS AND LOCATIONS:
Overall Officials: Hollie A Raynor, Ph.D, Study Director — The University of Tennessee, Knoxville; Susan B MacArthur, B.S., Principal Investigator — The University of Tennessee, Knoxville
Locations (1):
- The Early Learning Center, Knoxville, Tennessee, United States